CLINICAL TRIAL: NCT00007124
Title: A Trial of Ketogenic Diet in Lafora Disease
Brief Title: Ketogenic Diet in Lafora Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010042; 01-N-0042
Record Dates: First submitted 2000-12-07; First posted 2000-12-08 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-11

CONDITIONS: Lafora Disease
Keywords: Myoclonus; Epilepsy; Dementia; Polyglucosan; Insulin; Lafora Disease; Restrictive Carbohydrate Diet
MeSH Terms: conditions — Lafora Disease; Myoclonus; Epilepsy; Dementia; Insulin Resistance

SUMMARY:
This study will examine the effect of a restricted-carbohydrate diet (ketogenic diet) on Lafora disease-a severe neurological disease in which brain cells die because of abnormal accumulation of glucose (a type of sugar). Patients with Lafora disease have rapid neurological deterioration with myoclonus (brief muscle jerks), seizures and mental decline. At present there is no treatment to halt disease progression.

Patients 10 years of age and older with relatively advanced Lafora disease may be eligible for this study. Participants will be admitted to the Clinical Center for the first 4 weeks of this 6-month study for baseline testing and to start the ketogenic diet. They will have a complete medical history and physical examination, plus a detailed neurological examination and blood and urine tests. Procedures include:

* Magnetic resonance imaging (MRI) brain scans to provide information about brain chemistry
* Lumbar puncture (spinal tap) to analyze chemicals in cerebrospinal fluid
* Metabolic and endocrinological tests, including a glucose tolerance test, to evaluate the body's response to a large intake of oral glucose
* Standard neuropsychological tests
* Magnetic resonance spectroscopy of the brain and muscle
* Electroencephalography (EEG) to measure brain wave activity
* Electromyography (EMG) to measure muscle activity
* Evoked potentials (SEP and VEP) to study brain responses to mild electric or visual stimulation.

Transcranial magnetic stimulation (magnetic stimulation of the brain) may also be done to study the function of the brain cortex (outer nervous tissue of the brain) and the effects of treatment on brain excitability.

The ketogenic diet will begin after the tests are completed. The diet provides mainly fats to fuel the body, plus the recommended amount of protein and minimum carbohydrate. Vitamin and mineral supplements are provided to meet daily requirements. After 2 weeks on the diet, the patient will be discharged from the hospital and seen daily as an outpatient for another 1 to 2 weeks. During this time the patient or caregiver is trained in preparing the ketogenic diet, and then the patient is discharged to home. Throughout the study, disease symptoms will be assessed using standardized rating scales. Blood and urine tests will be done as needed, as will follow-up brain imaging, neuropsychological and neurophysiological evaluations.

A skin and/or muscle biopsy may be done at the first clinic visit to grow skin cells in culture and to analyze the skin and muscle under a microscope. The biopsy area is numbed with an anesthetic and a small piece of tissue is removed either with a needle, an instrument similar to a cookie-cutter or a knife. The skin cells may be used for metabolic studies and to obtain DNA for genetic testing.

At the end of the study, patients who responded well to the treatment with no significant adverse side effects may continue the diet for another 12 months. They will be followed at 3-month intervals to monitor side effects and treatment response.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the acute effect and potential disease modifying effects of a restrictive minimum carbohydrate diet (ketogenic diet) in patients with Lafora Disease. Untreated Lafora Disease is rapidly progressive to death over about 10 years. In an open label, proof-of-principle clinical trial, the efficacy of the ketogenic diet will be assessed through the use of validated clinical scales, as well as surrogate neurophysiological and biochemical measures. Safety will be monitored by means of frequent clinical evaluations and laboratory tests.

ELIGIBILITY:
Males and females older than 10 years will be eligible for this study. Younger children may not be sufficiently cooperative.

Women of child-bearing age must be using adequate contraceptive method for at least one month prior to and during participation in the study.

All will carry the diagnosis of Lafora disease based on the presence of characteristic clinical history and neurological findings.

All will have a relatively advanced disease with at least one of the three cardinal neurological manifestations: myoclonus, epilepsy and cognitive decline.

All patients will have histological or (preferable) genetic confirmation of diagnosis.

All patients will also be on stable doses of concomitant medications for at least 2 weeks prior to the onset of the study.

Patients must not have the presence or history of any medical condition that can reasonably be expected to subject the patient to unwarranted risk.

Patients must have no clinically significant laboratory abnormality that can reasonably be expected to subject the patient to unwarranted risk.

Patients must not have contraindications to the use of ketogenic diet: carnitine deficiency, organic acidurias, defects in beta-oxidation, clinically significant nephrolithiasis, and those who are immunosuppressed .

Pregnant women will be excluded. Those not practicing effective means of birth control will be excluded since the influence of this investigational therapy on the unborn child and reproductive organs is unknown. Urine pregnancy test will be performed on women of childbearing age.

Forbidden medications:

No significant interactions are generally expected between therapy with ketogenic diet and other concomitant medications. However, those carbohydrate-containing drug preparations which may interfere with the achievement of persistent ketosis, will be avoided as possible. Moreover, in case of unexpected hospital visits requiring IV fluids, patients and their parents will be asked to advise the treating medical staff on the need to avoid the use of dextrose-containing solutions, to minimize risks of iatrogenic seizures.

Anticonvulsant medications, in general, do not negatively interact with the ketogenic diet, but concomitant use of drugs such as Topiramate (sometimes associated with nephrolithiasis) will be avoided as possible.

As mentioned earlier, doses of VPA, commonly used in patients with myoclonic epilepsy, will be decreased by 25%, as KD may significantly elevate serum plasma levels of VPA.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15
Dates: Start 2000-12; Study Completion 2002-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Elliott EJ, Talbot IC, Pye IF, Hodges S, Swift PG, Tanner MS. Lafora disease: a progressive myoclonus epilepsy. J Paediatr Child Health. 1992 Dec;28(6):455-8. doi: 10.1111/j.1440-1754.1992.tb02717.x. PMID 1466943
- [Background] Berkovic SF, So NK, Andermann F. Progressive myoclonus epilepsies: clinical and neurophysiological diagnosis. J Clin Neurophysiol. 1991 Jul;8(3):261-74. PMID 1918332
- [Background] Federico A, D'Amore I, Palladini G, Medolago-Albani L, Guazzi GC, Tomaccini D. Lafora's disease. Clinical, histological ultrastructural and biochemical study. Acta Neurol (Napoli). 1980 Dec;2(6):466-75. No abstract available. PMID 6457518